CLINICAL TRIAL: NCT05849454
Title: Messy Memories: A Mobile Application Exposure Therapy Intervention to Reduce Psychological Distress and Improve Health Behaviors Following Critical Illness
Brief Title: Messy Memories: Mobile Application Therapy Following Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nadia A. Liyanage-Don, Assistant Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU1653; 5P30AG064198-04 (NIH)
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Psychological Distress; Health Behavior
Keywords: Critical Illness; Psychological Distress; Health Behavior; Post Traumatic Stress Disorder; Exposure Therapy; Intervention; Mental Disorders; Feasibility; Acceptability; Mobile Application; Intensive Care Unit; Trauma; Adherence
MeSH Terms: conditions — Critical Illness; Health Behavior; Stress Disorders, Post-Traumatic; Mental Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Messy Memories Intervention (Experimental): All participants enrolled in the study will be assigned to the experimental arm and participate in the Messy Memories intervention.
  Interventions: Device: Messy Memories Intervention

INTERVENTIONS:
Device: Messy Memories Intervention — Messy Memories is a mobile application that allows users to self-administer exposure therapy techniques outside of the traditional psychotherapy context. Participants are asked to audio record a difficult ("messy") memory, including what they did, felt, thought, smelled, saw, etc. They are then asked questions about what it was like to re-experience the memory, such as what emotions were elicited (e.g., sadness, anger, fear). Next, participants are asked to process what the memory means to them. They are then instructed to listen to their recording as often as they like, until the memory becomes easier to re-experience. They respond to processing questions each time they listen to their prior difficult memory.

SUMMARY:
The overall goal of this study is to determine whether English-speaking adults who were discharged from an intensive care unit (ICU) at least one month ago and have some level of distress related to their ICU experience will be interested in, willing to use, and satisfied with a new mobile application (app) designed to help the user process a difficult memory. Participants must have internet access and a smartphone in order to use the app. The goal of the app is to help reduce the psychological distress associated with a memory by processing that memory at one's own pace with app guidance. Participants will be asked to use the app for 6 weeks at least 3 times a week for 30 or more minutes at a time. Participants will also be asked to complete questionnaires over a 12-week period.

The investigators aim to test how possible and realistic it is for people who were hospitalized with a critical illness to voluntarily use this app to process relevant distressing memories of their hospitalization. The investigators hope that these results will inform the design of a larger trial that will be able to test if this app can reduce distress in this patient population, as the app may offer affordable and accessible help for some patients experiencing illness-related distress.

DETAILED DESCRIPTION:
Critical illness can be an incredibly traumatic experience, often involving treatment in the intensive care unit (ICU), intubation or other invasive medical procedures, altered levels of consciousness, inability to communicate, sensory and sleep deprivation, physical pain, and delirium. The cumulative physical and psychological stress associated with critical illness can be severe enough to induce clinically-significant symptoms of posttraumatic stress disorder (PTSD). Patients with PTSD symptoms related to prior traumatic medical events are more likely to engage in unhealthy behaviors, such as tobacco use, sedentary lifestyle, poor diet, and medication nonadherence.

Exposure therapy (ET) is considered the gold standard treatment for PTSD and involves repeated exposure to trauma-related stimuli leading to habituation of maladaptive emotional responses and an increased sense of control and self-competence. ET is highly effective for improving PTSD triggered by more typical forms of trauma, such as military combat or sexual assault, but less is known about the role of ET for reducing PTSD symptoms after critical illness.

The goal of this pilot study is to conduct preliminary testing of a newly developed mobile application (Messy Memories) that uses remotely delivered ET to reduce psychological distress and improve health behaviors in survivors of critical illness. The user is asked to audio record a traumatic or distressing memory and process what it feels like to re-experience the memory. Users can return to their recorded memory as often as they like until it becomes easier to re-experience.

The investigators will assess the feasibility and acceptability of recruiting and engaging critical illness survivors in the Messy Memories intervention. They will also explore the efficacy of the intervention for engaging the mechanistic target (PTSD symptoms) to reduce psychological distress. Additional outcomes will include reduction in other psychological symptoms (e.g., depression, anxiety) and improvement in health behaviors (e.g., sleep patterns, physical activity). The results of this study will form the basis of a future adequately powered randomized controlled trial testing whether the Messy Memories intervention can significantly reduce psychological distress and, in turn, improve behavioral outcomes among critical illness survivors.

Aim 1: Assess the feasibility of recruiting and engaging critical illness survivors in a mobile application-based exposure therapy intervention (Messy Memories). Hypothesis: The intervention will be feasible based on recruitment, retention, and completion rates of ≥70%.

Aim 2: Assess the acceptability of recruiting and engaging critical illness survivors in a mobile application-based exposure therapy intervention (Messy Memories). Hypothesis: The intervention will be acceptable based on participant satisfaction ratings of ≥70% and qualitative analysis of exit survey responses.

Aim 3 (exploratory): Assess engagement of the mechanistic target (PTSD symptoms) by the mobile application-based exposure therapy intervention (Messy Memories). Hypothesis: Participants will report improvement in PTSD symptoms, based on pre-/post-intervention decrease in scores on the PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5).

Participants will be asked to engage with the Messy Memories application at least 3 days a week for at least 30 minutes each day using their own mobile smartphone device. Participants may proceed through the modules of the application at their own pace and may return to any module as many times as they desire throughout the 6-week intervention period. Mechanistic target and clinical symptom assessments will occur at Week 0 (baseline), Week 3 (mid-intervention), Week 6 (end of intervention), and Week 12 (follow-up). All study procedures, including eligibility screening, consent process, outcome assessments, and exit surveys, will be conducted remotely via telephone or Zoom video conference.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Able to speak and write in English
* Previously admitted to an ICU
* Have internet access (e.g., Wi-Fi)
* Have access to an internet-equipped smartphone device (e.g., iPhone, Android)
* Meet a minimum threshold of psychological distress related to their prior critical illness as demonstrated by scoring ≥10 points on the PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5, see Measures section for a complete description).

Exclusion Criteria:

* ICU discharge occurred <30 days prior to the time of study enrollment
* Score <10 points on the PCL-5 during the initial eligibility screening
* Unable to comply with the protocol (either self-selected or indicating that s/he/they cannot complete all requested tasks) for reasons that include, but are not limited to, cognitive impairment (e.g., dementia), alcohol and/or substance abuse, or severe mental illness (e.g., schizophrenia).
* Unavailable for follow-up for reasons such as terminal illness and imminent plans to leave the United States (as this study may include migrant or mobile patients due to their citizenship and work issues).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Liyanage-Don, MD, MS, Principal Investigator — Columbia University; Ian Kronish, MD, MPH, Study Director — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ICU survivors were recruited nationwide between October 1, 2023 and May 31, 2024. The study was advertised to intensivists, post-ICU support groups, and ICU recovery clinics, as well as through online registries (e.g., RecruitMe, ResearchMatch, ClinicalTrials.gov), patient advocacy organizations (e.g., Sudden Cardiac Arrest Foundation), and relevant Facebook groups (e.g., ICU Survivor Support Group). IRB-approved flyers, emails, and presentations were used to promote the study.
Period: Overall Study
Arm/Group | Messy Memories Intervention
Started | 69
Screened Eligible for Study | 45
Signed Consent Form | 29
Completed Baseline Visit | 25
Completed 3-Week Visit | 22
Completed 6-Week Visit | 19
Completed 12-Week Visit | 20
Completed | 19
Not Completed | 50

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of the 29 participants who consented to study enrollment are reported below
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Region of Enrollment [Number; unit: Participants]
  United States | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Education [Count of Participants; unit: Participants]
  Trade/Vocational School | 1
  Some College | 9
  Associate's Degree | 2
  College Graduate | 10
  Graduate/Professional School | 7
Annual Household Income [Count of Participants; unit: Participants]
  <$10,000 | 2
  $10,000 - $24,999 | 2
  $25,000 - $49,999 | 4
  $50,000 - $74,999 | 5
  $75,000 - $99,999 | 10
  ≥$100,000 | 5
  Declined | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Screened Participants Who Screen Eligible for the Study
Description: This is designed to measure the feasibility of study recruitment
Time Frame: Baseline (pre-intervention)
Population: Because this was a feasibility study, we were interested in examining how many individuals needed to be screened to reach the target sample. Therefore, one of our primary outcome measures was the proportion of screened participants who screened eligible for the study. This would necessarily make the overall number of participants analyzed for this measure greater than the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 69
percentage of participants | 65.22 [53.62 to 75.36]

2. Primary Outcome: Percentage of Eligible Participants Who Enroll in the Study
Description: This is designed to measure the feasibility of study enrollment
Time Frame: Baseline (pre-intervention)
Population: Because this was a feasibility study, we were interested in examining how many individuals who screened eligible for the study would ultimately consent to study enrollment. Therefore, one of our primary outcome measures was the proportion of eligible participants who enrolled in the study. This would necessarily make the overall number of participants analyzed for this measure greater than the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 45
percentage of participants | 64.44 [51.11 to 77.78]

3. Primary Outcome: Percentage of Enrolled Participants Who Record a Memory in the Memory Processing Module
Description: This is designed to measure the feasibility of engaging with the intervention
Time Frame: End of 6-week intervention period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 29
percentage of participants | 65.52 [48.28 to 82.76]

4. Primary Outcome: Mean Number of Times That the Memory Processing Module is Accessed
Description: This is designed to measure the feasibility of engaging with the intervention. Of note, this outcome measure reflects the mean number of times per participant that the Memory Processing module was used to record a new memory or replay a previously recorded memory.
Time Frame: End of 6-week intervention period
Population: Not all participants who enrolled in the study engaged with the Messy Memories app, hence the difference between the number of participants analyzed here and the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Mean (Standard Deviation); unit: access per participant
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
access per participant | 5.00 (3.25)

5. Primary Outcome: Mean Duration of Time Spent Using the Memory Processing Module
Description: This is designed to measure the feasibility of engaging with the intervention
Time Frame: End of 6-week intervention period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
minutes | 57.37 (53.10)

6. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Feasibility
Description: Intervention feasibility will be measured with the Feasibility of Intervention Measure (FIM). The FIM is a 4-item questionnaire answered on a 5-point Likert scale (1 = completely disagree, 5 = completely agree). Responses to each item are averaged to obtain an overall score ranging from 1-5, with higher scores indicating a better outcome. Feasibility is defined as a score ≥4.
Time Frame: End of 6-week intervention period
Population: Not all participants who enrolled in the study completed the 6-week (post-intervention) visit during which the FIM was administered, hence the difference between the number of participants analyzed here and the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
percentage of participants | 78.95 [56.67 to 91.49]

7. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Acceptability
Description: Intervention acceptability will be measured with the Acceptability of Intervention Measure (AIM). The AIM is a 4-item questionnaire answered on a 5-point Likert scale (1 = completely disagree, 5 = completely agree). Responses to each item are averaged to obtain an overall score ranging from 1-5, with higher scores indicating a better outcome. Acceptability is defined as a score ≥4.
Time Frame: End of 6-week intervention period
Population: Not all participants who enrolled in the study completed the 6-week (post-intervention) visit during which the AIM was administered, hence the difference between the number of participants analyzed here and the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
percentage of participants | 73.68 [51.21 to 88.19]

8. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Appropriateness for Improving Psychological Distress
Description: Intervention appropriateness will be measured with the Intervention Appropriateness Measure (IAM). The IAM is a 4-item questionnaire answered on a 5-point Likert scale (1 = completely disagree, 5 = completely agree). Responses to each item are averaged to obtain an overall score ranging from 1-5, with higher scores indicating a better outcome. Appropriateness is defined as a score ≥4.
Time Frame: End of 6-week intervention period
Population: Not all participants who enrolled in the study completed the 6-week (post-intervention) visit during which the IAM was administered, hence the difference between the number of participants analyzed here and the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
percentage of participants | 68.42 [46.01 to 84.64]

9. Primary Outcome: Percentage of Participants Who Report Total Scores ≥68 for Their Final Rating of the Intervention's Usability
Description: Intervention usability will be measured with the System Usability Scale (SUS). The SUS is a 10-item questionnaire answered on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Scores range from 0-100, with higher scores indicating a better outcome. Usability is defined as a score ≥68.
Time Frame: End of 6-week intervention period
Population: Not all participants who enrolled in the study completed the 6-week (post-intervention) visit during which the SUS was administered, hence the difference between the number of participants analyzed here and the number of participants assigned to the arms or groups in the Participant Flow.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 19
percentage of participants | 73.68 [51.21 to 88.19]

10. Secondary Outcome: Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5) Score
Description: Post-traumatic stress symptoms triggered by the prior critical illness and ICU hospitalization will be assessed using the Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5). Participants are asked to rate how bothered they have been by each of 20 items in the past month on a 5-point Likert scale (0 = not at all, 4 = extremely). Items are summed to provide a total severity score ranging from 0-80, with higher scores indicating greater PTSD symptoms. A cut-point score ≥33 is considered positive for post-traumatic stress symptoms in civilian/primary care populations.
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: mean score on PCL-5 at 12 weeks
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
mean score on PCL-5 at 12 weeks | 21.40 (16.09)

11. Secondary Outcome: Patient Health Questionnaire (PHQ-8) Score
Description: Depression will be assessed using the Patient Health Questionnaire (PHQ-8). Participants are asked to rate how bothered they have been by each of 8 items in the past two weeks on a 4-point Likert scale (0 = not at all, 3 = nearly every day). Items are summed to provide a total severity score ranging from 0-24, with higher scores indicating greater depression. A cut-point score ≥10 is considered positive for depression.
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: mean score on PHQ-8 at 12 weeks
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
mean score on PHQ-8 at 12 weeks | 6.75 (5.24)

12. Secondary Outcome: Generalized Anxiety Disorder Scale (GAD-7) Score
Description: Anxiety will be assessed using the Generalized Anxiety Disorder Scale (GAD-7). Participants are asked to rate how bothered they have been by each of 7 items in the past two weeks on a 4-point Likert scale (0 = not at all, 3 = nearly every day). Items are summed to provide a total severity score ranging from 0-21, with higher scores indicating greater anxiety. A cut-point score ≥10 is considered positive for anxiety.
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: mean score on GAD-7 at 12 weeks
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
mean score on GAD-7 at 12 weeks | 5.25 (4.51)

13. Secondary Outcome: Anxiety Sensitivity Index (ASI) Score
Description: Anxiety sensitivity will be assessed using the Anxiety Sensitivity Index (ASI). Participants are asked to rate each of 16 items specifying different concerns someone could have regarding their anxiety on a 5-point Likert scale (0 = very little, 4 = very much). Items are summed to provide a total severity score ranging from 0-48, with higher scores indicating greater anxiety sensitivity. A cut-point score ≥17 is considered positive for anxiety sensitivity.
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: mean score on ASI at 12 weeks
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
mean score on ASI at 12 weeks | 23.65 (12.56)

14. Secondary Outcome: International Physical Activity Questionnaire (IPAQ) Score
Description: The 7-item subscale of the International Physical Activity Questionnaire (IPAQ) will be used to measure physical activity. Participants are asked to self-report the intensity, frequency, and duration of physical activity performed over the last 7 days. Responses are converted to metabolic equivalent of task (MET) minutes/week. Scores range from 0 MET minutes/week to 19,782 MET minutes/week, with higher scores indicating greater physical activity. There are no official cut-points for this subscale, but it may be dichotomized as "sufficient physical activity" (≥500 MET minutes/week) vs "insufficient physical activity" (<500 MET minutes/week).
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: mean score on IPAQ at 12 weeks
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
mean score on IPAQ at 12 weeks | 3772 (4179)

15. Secondary Outcome: Number of Hours of Sleep
Description: Participants will be asked "During the past month, how many hours of actual sleep did you get at night (this may be different than the number of hours you spent in bed)?" Responses are given in number of hours and range from 0 to >10, with higher values indicating greater hours of sleep. There are no official cut-points for this item, but it may be dichotomized as "short sleep duration" (< 7 hours of sleep) vs "not short sleep duration" (≥7 hours of sleep).
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: hours of sleep per night
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
hours of sleep per night | 6.75 (1.80)

16. Secondary Outcome: Self-reported Use of Sleep Medication
Description: Participants will be asked "During the past month, how often have you taken medicine to help you sleep (prescribed or 'over the counter')?" Responses are given on a 4-point Likert scale (0 = not during the past month, 1 = less than once a week, 2 = once or twice a week, 3 = three of more times a week), with higher values indicating greater medication use. There are no official cut-points for this item, but it may be dichotomized as "no habitual use of sleep medication" (score of 0 or 1) vs "at least some use of sleep medication" (score of 2 or 3).
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
score on a scale | 0.85 (1.18)

17. Secondary Outcome: Rating of Sleep Quality
Description: Participants will be asked "During the past month, how would you rate your sleep quality overall?" Responses are given on a 4-point Likert scale (0 = very good, 1 = fairly good, 2 = fairly bad, 3 = very bad), with higher values indicating worse sleep quality. There are no official cut-points for this item, but it may be dichotomized as "good quality sleep" (score of 0 or 1) vs "bad quality sleep" (score of 2 or 3).
Time Frame: 12 weeks
Population: Data are reported for the 20 participants who completed the 12-week visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Messy Memories Intervention
Number analyzed (Participants) | 20
score on a scale | 0.85 (0.88)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 weeks
Arm/Group | Messy Memories Intervention
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Limitations include inability to confirm self-reported ICU history and potential for imposter participants due to remote nature of the study. Participants received technical/onboarding support that is not typical of many apps, which may have influenced engagement. The app's availability in English only and the need for an internet-accessible smartphone limits generalizability. Finally, the small sample and lack of control group constrain our ability to draw strong conclusions about efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT05849454/Prot_SAP_000.pdf